CLINICAL TRIAL: NCT00018382
Title: Insulin, Neurogenetics and Memory in Alzheimer's Disease: A Novel Therapeutic Approach
Brief Title: Insulin, Neurogenetics and Memory in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: AGCG-012-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
This study examines the use of insulin-sensitizing compounds, as therapeutic agents for cognitive impairment in Alzheimer's disease.

ELIGIBILITY:
Men and women with mild Alzheimer's Disease without serious medical or psychiatric comorbid conditions.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kahn, M.D.; Sanjay Asthana, M.D.; Alfred Fujimoto, M.D.
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States